CLINICAL TRIAL: NCT05219006
Title: Ketogenic Diet Effects on the Frequency of Non Epileptic Seizures in Patients With Dissociative Neurological Symptom Disorder: a Pilot Study
Brief Title: Ketogenic Diet Effects on the Frequency of Non Epileptic Seizures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez (Other)
Responsible Party: Principal Investigator, Edgar Daniel Crail Melendez, MS, El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8/21
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Non Epileptic Seizures; Functional Neurological Symptom Disorder; Conversion Disorder; Ketogenic Dieting
MeSH Terms: conditions — Seizures; Conversion Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketogenic dieting + conventional treatment (Experimental): Nutrition team will help patients implement an Atkins-type ketogenic diet. The diet should be continued for at least 6 weeks. They will be able to continue with the pharmacological-based treatment but without any changes having been made in the last 6 weeks or during the time they are in the study. To ensure adherence to the diet, urine ketones will be determined twice a week.
  Interventions: Dietary Supplement: ketogenic dieting
- Healthy dieting + conventional treatment (Active Comparator): In addition to their basic (pharmacological) treatment, the nutrition team will help them implement a low-calorie, non-ketogenic diet. The presence of ketones will also be determined in urine to avoid bias
  Interventions: Dietary Supplement: healthy dieting

INTERVENTIONS:
Dietary Supplement: ketogenic dieting — Atkins modified diet: 1.2-1.5 g/kg/day of protein with a ratio 1:1 (fat: carbohydrate + protein)
  Arms: ketogenic dieting + conventional treatment
Dietary Supplement: healthy dieting — Normocaloric diet established by a nutritionist. 1.2-1.5 g/kg/day of protein with a maximum contribution of 50 % carbohydrates of the total calorie intake eliminating industrialized food.
  Arms: Healthy dieting + conventional treatment

SUMMARY:
The objective of this study is to determine the effects of the ketogenic diet on the frequency of non-epileptic seizures in patients with functional neurological symptoms disorder compared to a healthy diet.

DETAILED DESCRIPTION:
This study consists of a open label randomized controlled clinical trial comprised of 20 patients with diagnosis of functional neurological symptom disorder with non epileptic seizures distributed in 2 arms of 10 patients each.

Patients will be randomly assigned to one of the groups. Both groups will be receiving treatment as usual (SSRI and/or psychotherapy). One group will be assigned a ketogenic diet while the other will be assigned a healthy diet, both supervised by a team of nutritionists. Patients will be evaluated every 2 weeks until reaching 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a record at the institute and who have a diagnosis of a dissociative neurological symptom disorder with non-epileptic seizures with a certainty of at least clinically established who have a monthly seizure frequency greater than 3.
* Patients with the characteristics described above with comorbid epilepsy but who have not presented epileptic seizures in the last month.
* Patients with the aforementioned characteristics and who give their informed consent in writing to participate in the study.
* Patients who, once the diet has been explained to them, consider it feasible to implement it at least for the follow-up time.

Exclusion Criteria:

* Patients with metabolic or hemodynamic instability, liver failure, inability to tolerate the oral route, acute pancreatitis or pregnancy due to the possible teratogenic effect that has not yet been elucidated.
* Patients with metabolic disorders such as primary carnitine deficiency, palmitoyltransferase carnitine I or II deficiency, carnitine translocase deficiency, beta oxidation defects, pyruvate carboxylase deficiency, porphyria and other fatty acid transport and oxidation disorders.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-07-02 (Actual)

PRIMARY OUTCOMES:
non epileptic seizure frequency | 2 weeks
  number of non epileptic seizures the patient reports on a written crisis record with the aid of a caregiver if necessary

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Crail Meléndez, MS, Principal Investigator — El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez
Locations (1):
- Instituto Nacional de Neurologia Y Neurocirugia Mvs, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Popkirov S, Asadi-Pooya AA, Duncan R, Gigineishvili D, Hingray C, Miguel Kanner A, LaFrance WC Jr, Pretorius C, Reuber M. The aetiology of psychogenic non-epileptic seizures: risk factors and comorbidities. Epileptic Disord. 2019 Dec 1;21(6):529-547. doi: 10.1684/epd.2019.1107. PMID 31843732
- [Background] Avbersek A, Sisodiya S. Does the primary literature provide support for clinical signs used to distinguish psychogenic nonepileptic seizures from epileptic seizures? J Neurol Neurosurg Psychiatry. 2010 Jul;81(7):719-25. doi: 10.1136/jnnp.2009.197996. PMID 20581136
- [Background] Kanemoto K, LaFrance WC Jr, Duncan R, Gigineishvili D, Park SP, Tadokoro Y, Ikeda H, Paul R, Zhou D, Taniguchi G, Kerr M, Oshima T, Jin K, Reuber M. PNES around the world: Where we are now and how we can close the diagnosis and treatment gaps-an ILAE PNES Task Force report. Epilepsia Open. 2017 Jun 23;2(3):307-316. doi: 10.1002/epi4.12060. eCollection 2017 Sep. PMID 29588959
- [Background] Hingray C, Maillard L, Hubsch C, Vignal JP, Bourgognon F, Laprevote V, Lerond J, Vespignani H, Schwan R. Psychogenic nonepileptic seizures: characterization of two distinct patient profiles on the basis of trauma history. Epilepsy Behav. 2011 Nov;22(3):532-6. doi: 10.1016/j.yebeh.2011.08.015. Epub 2011 Oct 1. PMID 21962755
- [Background] Sigurdardottir KR, Olafsson E. Incidence of psychogenic seizures in adults: a population-based study in Iceland. Epilepsia. 1998 Jul;39(7):749-52. doi: 10.1111/j.1528-1157.1998.tb01161.x. PMID 9670904
- [Background] Stone J, Carson A, Duncan R, Roberts R, Warlow C, Hibberd C, Coleman R, Cull R, Murray G, Pelosi A, Cavanagh J, Matthews K, Goldbeck R, Smyth R, Walker J, Sharpe M. Who is referred to neurology clinics?--the diagnoses made in 3781 new patients. Clin Neurol Neurosurg. 2010 Nov;112(9):747-51. doi: 10.1016/j.clineuro.2010.05.011. Epub 2010 Jun 19. PMID 20646830
- [Background] Benbadis SR, Allen Hauser W. An estimate of the prevalence of psychogenic non-epileptic seizures. Seizure. 2000 Jun;9(4):280-1. doi: 10.1053/seiz.2000.0409. PMID 10880289
- [Background] Asadi-Pooya AA, Sperling MR. Epidemiology of psychogenic nonepileptic seizures. Epilepsy Behav. 2015 May;46:60-5. doi: 10.1016/j.yebeh.2015.03.015. Epub 2015 Apr 14. PMID 25882323
- [Background] Goldstein LH, Robinson EJ, Reuber M, Chalder T, Callaghan H, Eastwood C, Landau S, McCrone P, Medford N, Mellers JDC, Moore M, Mosweu I, Murray J, Perdue I, Pilecka I, Richardson MP, Carson A, Stone J; CODES Study Group. Characteristics of 698 patients with dissociative seizures: A UK multicenter study. Epilepsia. 2019 Nov;60(11):2182-2193. doi: 10.1111/epi.16350. Epub 2019 Oct 13. PMID 31608436
- [Background] Duncan R, Oto M, Wainman-Lefley J. Mortality in a cohort of patients with psychogenic non-epileptic seizures. J Neurol Neurosurg Psychiatry. 2012 Jul;83(7):761-2. doi: 10.1136/jnnp-2012-302900. PMID 22665451
- [Background] LaFrance Jr W, Bjørnaes H. Designing treatment plans based on etiology of psychogenic nonepileptic seizures. Gates and Rowan's nonepilepfic seizures. 2010:266-80.
- [Background] Brown RJ, Reuber M. Towards an integrative theory of psychogenic non-epileptic seizures (PNES). Clin Psychol Rev. 2016 Jul;47:55-70. doi: 10.1016/j.cpr.2016.06.003. Epub 2016 Jun 17. No abstract available. PMID 27340856
- [Background] Reuber M, Brown RJ. Understanding psychogenic nonepileptic seizures-Phenomenology, semiology and the Integrative Cognitive Model. Seizure. 2017 Jan;44:199-205. doi: 10.1016/j.seizure.2016.10.029. Epub 2016 Nov 15. PMID 27988107
- [Background] Devinsky O, Gazzola D, LaFrance WC Jr. Differentiating between nonepileptic and epileptic seizures. Nat Rev Neurol. 2011 Apr;7(4):210-20. doi: 10.1038/nrneurol.2011.24. Epub 2011 Mar 8. PMID 21386814
- [Background] Brigo F, Nardone R, Ausserer H, Storti M, Tezzon F, Manganotti P, Bongiovanni LG. The diagnostic value of urinary incontinence in the differential diagnosis of seizures. Seizure. 2013 Mar;22(2):85-90. doi: 10.1016/j.seizure.2012.10.011. Epub 2012 Nov 9. PMID 23142708
- [Background] Syed TU, LaFrance WC Jr, Kahriman ES, Hasan SN, Rajasekaran V, Gulati D, Borad S, Shahid A, Fernandez-Baca G, Garcia N, Pawlowski M, Loddenkemper T, Amina S, Koubeissi MZ. Can semiology predict psychogenic nonepileptic seizures? A prospective study. Ann Neurol. 2011 Jun;69(6):997-1004. doi: 10.1002/ana.22345. Epub 2011 Mar 17. PMID 21437930
- [Background] Perez DL, LaFrance WC Jr. Nonepileptic seizures: an updated review. CNS Spectr. 2016 Jun;21(3):239-46. doi: 10.1017/S109285291600002X. Epub 2016 Mar 21. PMID 26996600
- [Background] LaFrance WC Jr, Baker GA, Duncan R, Goldstein LH, Reuber M. Minimum requirements for the diagnosis of psychogenic nonepileptic seizures: a staged approach: a report from the International League Against Epilepsy Nonepileptic Seizures Task Force. Epilepsia. 2013 Nov;54(11):2005-18. doi: 10.1111/epi.12356. Epub 2013 Sep 20. PMID 24111933
- [Background] Dixit R, Popescu A, Bagic A, Ghearing G, Hendrickson R. Medical comorbidities in patients with psychogenic nonepileptic spells (PNES) referred for video-EEG monitoring. Epilepsy Behav. 2013 Aug;28(2):137-40. doi: 10.1016/j.yebeh.2013.05.004. Epub 2013 Jun 5. PMID 23747495
- [Background] Duncan R, Oto M. Predictors of antecedent factors in psychogenic nonepileptic attacks: multivariate analysis. Neurology. 2008 Sep 23;71(13):1000-5. doi: 10.1212/01.wnl.0000326593.50863.21. PMID 18809836
- [Background] Perez DL, Dworetzky BA, Dickerson BC, Leung L, Cohn R, Baslet G, Silbersweig DA. An integrative neurocircuit perspective on psychogenic nonepileptic seizures and functional movement disorders: neural functional unawareness. Clin EEG Neurosci. 2015 Jan;46(1):4-15. doi: 10.1177/1550059414555905. Epub 2014 Nov 27. PMID 25432161
- [Background] Direk N, Kulaksizoglu IB, Alpay K, Gurses C. Using personality disorders to distinguish between patients with psychogenic nonepileptic seizures and those with epileptic seizures. Epilepsy Behav. 2012 Feb;23(2):138-41. doi: 10.1016/j.yebeh.2011.11.013. Epub 2012 Jan 10. PMID 22236571
- [Background] Myers L, Perrine K, Lancman M, Fleming M, Lancman M. Psychological trauma in patients with psychogenic nonepileptic seizures: trauma characteristics and those who develop PTSD. Epilepsy Behav. 2013 Jul;28(1):121-6. doi: 10.1016/j.yebeh.2013.03.033. Epub 2013 May 23. PMID 23708490
- [Background] Selkirk M, Duncan R, Oto M, Pelosi A. Clinical differences between patients with nonepileptic seizures who report antecedent sexual abuse and those who do not. Epilepsia. 2008 Aug;49(8):1446-50. doi: 10.1111/j.1528-1167.2008.01611.x. Epub 2008 Apr 10. PMID 18410361
- [Background] Goldstein LH, Chalder T, Chigwedere C, Khondoker MR, Moriarty J, Toone BK, Mellers JD. Cognitive-behavioral therapy for psychogenic nonepileptic seizures: a pilot RCT. Neurology. 2010 Jun 15;74(24):1986-94. doi: 10.1212/WNL.0b013e3181e39658. PMID 20548043
- [Background] LaFrance WC Jr, Keitner GI, Papandonatos GD, Blum AS, Machan JT, Ryan CE, Miller IW. Pilot pharmacologic randomized controlled trial for psychogenic nonepileptic seizures. Neurology. 2010 Sep 28;75(13):1166-73. doi: 10.1212/WNL.0b013e3181f4d5a9. Epub 2010 Aug 25. PMID 20739647
- [Background] Oto M, Espie CA, Duncan R. An exploratory randomized controlled trial of immediate versus delayed withdrawal of antiepileptic drugs in patients with psychogenic nonepileptic attacks (PNEAs). Epilepsia. 2010 Oct;51(10):1994-9. doi: 10.1111/j.1528-1167.2010.02696.x. Epub 2010 Aug 17. PMID 20726877
- [Background] Chen DK, Maheshwari A, Franks R, Trolley GC, Robinson JS, Hrachovy RA. Brief group psychoeducation for psychogenic nonepileptic seizures: a neurologist-initiated program in an epilepsy center. Epilepsia. 2014 Jan;55(1):156-66. doi: 10.1111/epi.12481. Epub 2013 Dec 20. PMID 24446955
- [Background] LaFrance WC Jr, Baird GL, Barry JJ, Blum AS, Frank Webb A, Keitner GI, Machan JT, Miller I, Szaflarski JP; NES Treatment Trial (NEST-T) Consortium. Multicenter pilot treatment trial for psychogenic nonepileptic seizures: a randomized clinical trial. JAMA Psychiatry. 2014 Sep;71(9):997-1005. doi: 10.1001/jamapsychiatry.2014.817. PMID 24989152
- [Background] Hipócrates. On the Sacred Disease. 400BC.
- [Background] Williams TJ, Cervenka MC. The role for ketogenic diets in epilepsy and status epilepticus in adults. Clin Neurophysiol Pract. 2017 Jul 1;2:154-160. doi: 10.1016/j.cnp.2017.06.001. eCollection 2017. PMID 30214989
- [Background] Cervenka MC, Kossoff EH. Dietary treatment of intractable epilepsy. Continuum (Minneap Minn). 2013 Jun;19(3 Epilepsy):756-66. doi: 10.1212/01.CON.0000431396.23852.56. PMID 23739109
- [Background] McNally MA, Hartman AL. Ketone bodies in epilepsy. J Neurochem. 2012 Apr;121(1):28-35. doi: 10.1111/j.1471-4159.2012.07670.x. Epub 2012 Feb 7. PMID 22268909
- [Background] Zupec-Kania BA, Spellman E. An overview of the ketogenic diet for pediatric epilepsy. Nutr Clin Pract. 2008 Dec-2009 Jan;23(6):589-96. doi: 10.1177/0884533608326138. PMID 19033218
- [Background] Klein P, Tyrlikova I, Mathews GC. Dietary treatment in adults with refractory epilepsy: a review. Neurology. 2014 Nov 18;83(21):1978-85. doi: 10.1212/WNL.0000000000001004. Epub 2014 Oct 29. PMID 25355830
- [Background] Payne NE, Cross JH, Sander JW, Sisodiya SM. The ketogenic and related diets in adolescents and adults--a review. Epilepsia. 2011 Nov;52(11):1941-8. doi: 10.1111/j.1528-1167.2011.03287.x. Epub 2011 Oct 17. PMID 22004525
- [Background] Muzykewicz DA, Lyczkowski DA, Memon N, Conant KD, Pfeifer HH, Thiele EA. Efficacy, safety, and tolerability of the low glycemic index treatment in pediatric epilepsy. Epilepsia. 2009 May;50(5):1118-26. doi: 10.1111/j.1528-1167.2008.01959.x. Epub 2009 Feb 12. PMID 19220406
- [Background] Neal EG, Cross JH. Efficacy of dietary treatments for epilepsy. J Hum Nutr Diet. 2010 Apr;23(2):113-9. doi: 10.1111/j.1365-277X.2010.01043.x. PMID 20487176
- [Background] Coppola G, D'Aniello A, Messana T, Di Pasquale F, della Corte R, Pascotto A, Verrotti A. Low glycemic index diet in children and young adults with refractory epilepsy: first Italian experience. Seizure. 2011 Sep;20(7):526-8. doi: 10.1016/j.seizure.2011.03.008. Epub 2011 Apr 13. PMID 21489826
- [Background] Pfeifer HH, Thiele EA. Low-glycemic-index treatment: a liberalized ketogenic diet for treatment of intractable epilepsy. Neurology. 2005 Dec 13;65(11):1810-2. doi: 10.1212/01.wnl.0000187071.24292.9e. PMID 16344529
- [Background] Kossoff EH, Cervenka MC, Henry BJ, Haney CA, Turner Z. A decade of the modified Atkins diet (2003-2013): Results, insights, and future directions. Epilepsy Behav. 2013 Dec;29(3):437-42. doi: 10.1016/j.yebeh.2013.09.032. PMID 24386671
- [Background] Lambrechts DA, Wielders LH, Aldenkamp AP, Kessels FG, de Kinderen RJ, Majoie MJ. The ketogenic diet as a treatment option in adults with chronic refractory epilepsy: efficacy and tolerability in clinical practice. Epilepsy Behav. 2012 Mar;23(3):310-4. doi: 10.1016/j.yebeh.2012.01.002. Epub 2012 Feb 25. PMID 22366051
- [Background] Smith M, Politzer N, Macgarvie D, McAndrews MP, Del Campo M. Efficacy and tolerability of the modified Atkins diet in adults with pharmacoresistant epilepsy: a prospective observational study. Epilepsia. 2011 Apr;52(4):775-80. doi: 10.1111/j.1528-1167.2010.02941.x. Epub 2011 Jan 26. PMID 21269295
- [Background] Trauner DA. Medium-chain triglyceride (MCT) diet in intractable seizure disorders. Neurology. 1985 Feb;35(2):237-8. doi: 10.1212/wnl.35.2.237. PMID 3969213
- [Background] Kossoff EH, Zupec-Kania BA, Amark PE, Ballaban-Gil KR, Christina Bergqvist AG, Blackford R, Buchhalter JR, Caraballo RH, Helen Cross J, Dahlin MG, Donner EJ, Klepper J, Jehle RS, Kim HD, Christiana Liu YM, Nation J, Nordli DR Jr, Pfeifer HH, Rho JM, Stafstrom CE, Thiele EA, Turner Z, Wirrell EC, Wheless JW, Veggiotti P, Vining EP; Charlie Foundation, Practice Committee of the Child Neurology Society; Practice Committee of the Child Neurology Society; International Ketogenic Diet Study Group. Optimal clinical management of children receiving the ketogenic diet: recommendations of the International Ketogenic Diet Study Group. Epilepsia. 2009 Feb;50(2):304-17. doi: 10.1111/j.1528-1167.2008.01765.x. Epub 2008 Sep 23. PMID 18823325
- [Background] Ye F, Li XJ, Jiang WL, Sun HB, Liu J. Efficacy of and patient compliance with a ketogenic diet in adults with intractable epilepsy: a meta-analysis. J Clin Neurol. 2015 Jan;11(1):26-31. doi: 10.3988/jcn.2015.11.1.26. Epub 2015 Jan 2. PMID 25628734
- [Background] Kverneland M, Selmer KK, Nakken KO, Iversen PO, Tauboll E. A prospective study of the modified Atkins diet for adults with idiopathic generalized epilepsy. Epilepsy Behav. 2015 Dec;53:197-201. doi: 10.1016/j.yebeh.2015.10.021. Epub 2015 Nov 14. PMID 26588588
- [Background] Schoeler NE, Wood S, Aldridge V, Sander JW, Cross JH, Sisodiya SM. Ketogenic dietary therapies for adults with epilepsy: feasibility and classification of response. Epilepsy Behav. 2014 Aug;37:77-81. doi: 10.1016/j.yebeh.2014.06.007. Epub 2014 Jul 8. PMID 25010319
- [Background] Cervenka MC, Henry BJ, Felton EA, Patton K, Kossoff EH. Establishing an Adult Epilepsy Diet Center: Experience, efficacy and challenges. Epilepsy Behav. 2016 May;58:61-8. doi: 10.1016/j.yebeh.2016.02.038. Epub 2016 Apr 6. PMID 27060389
- [Background] Johnson E, Cervenka M. Dietary therapy in adults: history, demand, and results. Ketogenic Diet and Metabolic Therapies: Expanded Roles in Health and Disease: Oxford University Press, New York; 2017. p. 16-25.
- [Background] Carrette E, Vonck K, de Herdt V, Dewaele I, Raedt R, Goossens L, Van Zandijcke M, Wadman W, Thadani V, Boon P. A pilot trial with modified Atkins' diet in adult patients with refractory epilepsy. Clin Neurol Neurosurg. 2008 Sep;110(8):797-803. doi: 10.1016/j.clineuro.2008.05.003. Epub 2008 Jun 24. PMID 18572306
- [Background] Hocker SE, Britton JW, Mandrekar JN, Wijdicks EF, Rabinstein AA. Predictors of outcome in refractory status epilepticus. JAMA Neurol. 2013 Jan;70(1):72-7. doi: 10.1001/jamaneurol.2013.578. PMID 23318514
- [Background] Olson CA, Vuong HE, Yano JM, Liang QY, Nusbaum DJ, Hsiao EY. The Gut Microbiota Mediates the Anti-Seizure Effects of the Ketogenic Diet. Cell. 2018 Jun 14;173(7):1728-1741.e13. doi: 10.1016/j.cell.2018.04.027. Epub 2018 May 24. PMID 29804833
- [Background] Kossoff EH, Al-Macki N, Cervenka MC, Kim HD, Liao J, Megaw K, Nathan JK, Raimann X, Rivera R, Wiemer-Kruel A, Williams E, Zupec-Kania BA. What are the minimum requirements for ketogenic diet services in resource-limited regions? Recommendations from the International League Against Epilepsy Task Force for Dietary Therapy. Epilepsia. 2015 Sep;56(9):1337-42. doi: 10.1111/epi.13039. Epub 2015 May 29. PMID 26033161
- [Background] Sirven J, Whedon B, Caplan D, Liporace J, Glosser D, O'Dwyer J, Sperling MR. The ketogenic diet for intractable epilepsy in adults: preliminary results. Epilepsia. 1999 Dec;40(12):1721-6. doi: 10.1111/j.1528-1157.1999.tb01589.x. PMID 10612335
- [Background] Cervenka MC, Patton K, Eloyan A, Henry B, Kossoff EH. The impact of the modified Atkins diet on lipid profiles in adults with epilepsy. Nutr Neurosci. 2016;19(3):131-7. doi: 10.1179/1476830514Y.0000000162. Epub 2014 Nov 10. PMID 25383724
- [Background] Klein P, Janousek J, Barber A, Weissberger R. Ketogenic diet treatment in adults with refractory epilepsy. Epilepsy Behav. 2010 Dec;19(4):575-9. doi: 10.1016/j.yebeh.2010.09.016. PMID 20937568
- [Background] Mosek A, Natour H, Neufeld MY, Shiff Y, Vaisman N. Ketogenic diet treatment in adults with refractory epilepsy: a prospective pilot study. Seizure. 2009 Jan;18(1):30-3. doi: 10.1016/j.seizure.2008.06.001. Epub 2008 Aug 3. PMID 18675556
- [Background] Paoli A, Rubini A, Volek JS, Grimaldi KA. Beyond weight loss: a review of the therapeutic uses of very-low-carbohydrate (ketogenic) diets. Eur J Clin Nutr. 2013 Aug;67(8):789-96. doi: 10.1038/ejcn.2013.116. Epub 2013 Jun 26. PMID 23801097
- [Background] Sharman MJ, Kraemer WJ, Love DM, Avery NG, Gomez AL, Scheett TP, Volek JS. A ketogenic diet favorably affects serum biomarkers for cardiovascular disease in normal-weight men. J Nutr. 2002 Jul;132(7):1879-85. doi: 10.1093/jn/132.7.1879. PMID 12097663
- [Background] Kossoff EH, Rowley H, Sinha SR, Vining EP. A prospective study of the modified Atkins diet for intractable epilepsy in adults. Epilepsia. 2008 Feb;49(2):316-9. doi: 10.1111/j.1528-1167.2007.01256.x. Epub 2007 Oct 5. PMID 17919301
- [Background] Cervenka MC, Terao NN, Bosarge JL, Henry BJ, Klees AA, Morrison PF, Kossoff EH. E-mail management of the modified Atkins Diet for adults with epilepsy is feasible and effective. Epilepsia. 2012 Apr;53(4):728-32. doi: 10.1111/j.1528-1167.2012.03406.x. Epub 2012 Feb 14. PMID 22332768
- [Background] Rivera Espinoza Y. Microbiota intestinal: su importancia en la salud y los factores que la modifican. Lat Am J Clin Sci Med Technol. 2020;2(2):185-96.
- [Background] Wikberg C, Pettersson A, Westman J, Bjorkelund C, Petersson EL. Patients' perspectives on the use of the Montgomery-Asberg depression rating scale self-assessment version in primary care. Scand J Prim Health Care. 2016 Dec;34(4):434-442. doi: 10.1080/02813432.2016.1248635. Epub 2016 Nov 2. PMID 27804312
- [Background] Vilagut G, Ferrer M, Rajmil L, Rebollo P, Permanyer-Miralda G, Quintana JM, Santed R, Valderas JM, Ribera A, Domingo-Salvany A, Alonso J. [The Spanish version of the Short Form 36 Health Survey: a decade of experience and new developments]. Gac Sanit. 2005 Mar-Apr;19(2):135-50. doi: 10.1157/13074369. Spanish. PMID 15860162